CLINICAL TRIAL: NCT00664781
Title: A Cancer Research UK Phase II Proof of Principle Trial of the Activity of the PARP-1 Inhibitor, AG-014699, in Known Carriers of a BRCA 1 or BRCA 2 Mutation With Locally Advanced or Metastatic Breast or Advanced Ovarian Cancer
Brief Title: Rucaparib(CO-338;Formally Called AG-014699 or PF-0136738) in Treating Patients With Locally Advanced or Metastatic Breast Cancer or Advanced Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000593558; CRUK-PH2-052; CRUK-PARP/BRCA; EU-20842; EUDRACT-2006-002348-27
Record Dates: First submitted 2008-04-22; First posted 2008-04-23 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: brca1 Mutation Carrier; brca2 Mutation Carrier; Breast Cancer; Ovarian Cancer
Keywords: stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent breast cancer; stage IV ovarian epithelial cancer; recurrent ovarian germ cell tumor; stage IV ovarian germ cell tumor; ovarian stromal cancer; ovarian sarcoma; BRCA1 mutation carrier; BRCA2 mutation carrier; stage IIIA ovarian epithelial cancer; stage IIIA ovarian germ cell tumor; stage IIIB ovarian epithelial cancer; stage IIIB ovarian germ cell tumor; stage IIIC ovarian epithelial cancer; stage IIIC ovarian germ cell tumor; ovarian papillary serous carcinoma
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — rucaparib; Blotting, Western; Immunohistochemistry; Chromatography, Liquid; Mass Spectrometry

INTERVENTIONS:
Drug: rucaparib (CO-338; formally AG-014699 or PF-01367338)
Genetic: protein expression analysis
Genetic: western blotting
Other: immunohistochemistry staining method
Other: liquid chromatography
Other: mass spectrometry
Other: pharmacological study

SUMMARY:
RATIONALE: rucaparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying the side effects and best dose of rucaparib and to see how well it works in treating patients with locally advanced or metastatic breast cancer or advanced ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assessment of Anti tumour activity to PARP-1 inhibitor rucaparib in patients with locally advanced or metastatic breast or advanced ovarian cancer shown to express the BRCA 1 or 2 mutations.
* To evaluate the toxicity of treatment with Rucaparib in these population's.

Secondary

* To evaluate the time to progression and overall survival in patients treated with this drug.
* To study pharmacokinetics of this drug in these patient populations.
* To evaluate the Poly(ADP-ribose) polymerase (PARP) activity in peripheral blood lymphocytes from BRCA 1 and 2 heterozygotic patients.
* To determine a tolerable and effective dosing regimen of the Rucaparib oral formulation.

OUTLINE: This is a dose-escalation study followed by an open label multicenter study. The study was originally set up with an IV formulation. An oral formulation of the PARP-1 inhibitor rucaparib will be used from now on. Patients are stratified according to tumor type (breast vs ovarian) and mutation status ( BRCA 1 vs BRCA 2). In addition, patient with high-grade serous ovarian cancer can be enrolled into Stage 1 of the study. All patients enrolled will receive PARP-1 inhibitor rucaparib oral formulation once daily for either 7, 14, or 21 days of each cycle, (two possible dosages for 21 days treatment). Treatment repeats every 21 days for 12 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve stable or responding disease may receive additional courses of treatment at the discretion of the chief investigator or Drug Development Office (DDO).

Patients undergo blood sample collection periodically for pharmacokinetic and pharmacodynamic studies. Samples are analyzed for tumor marker (CA 125 and/or CA 15.3) measurements, rucaparib plasma levels via liquid chromatography/mass spectrometry/mass spectrometry, PARP activity, and PARP protein expression via western blotting immunoassays. Paraffin embedded sections from original diagnostic biopsy are also collected and analyzed for PARP protein expression via immunohistochemical technique. Pleural and ascitic fluid may be collected and analyzed for DNA DS break repair proficiency via immunohistochemical technique. Some patients also undergo biopsy of tumors and samples are analyzed for BRCA 2 mutation as well as PARP activity via validated PARP immunoblotting assay.

After completion of study treatment, patients are followed for 28 days.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
INCLUSION CRITERIA

1. All stages of the study (IV and oral):

   Patients must be proven known carriers of a mutation of BRCA1 or BRCA2 or considered to be highly likely to be carriers of a BRCA1 or 2 mutation* (score of ≥ 20 as per Manchester criteria) and have histologically documented locally advanced or metastatic breast cancer or advanced ovarian cancer.

   *Patients considered highly likely to be carriers will be tested after consenting and a BRCA1 or 2 mutation must be confirmed for the patient to be eligible to receive treatment.

   Oral stage 1 only:

   In addition to the above, patients with high grade serous ovarian cancer with unknown BRCA status may be entered into oral stage 1.
2. Patients with ovarian cancer (including epithelial, fallopian tube cancer and primary peritoneal cancer) who have had no more than 5 prior chemotherapy regimens in the last 5 years. For the BRCA carriers > 2 months must have elapsed since their last treatment with a carboplatin- or cisplatin-containing regimen or for high grade serous ovarian cancer patients ≥ 6 months.
3. Patients with breast cancer who have had no more than 5 prior chemotherapy regimens in the last 5 years.
4. Measurable disease as measured by X-ray, computerised tomography (CT), or MRI scan as defined by RECIST criteria. These measurements must be done within 4 weeks of the patient going on study. Clinical measurements must be done within one week of the patient going on study. Patients with bone disease must have other measurable disease for evaluation. Previously irradiated lesions cannot be used for measurable disease.
5. Life expectancy of at least 12 weeks
6. World Health Organisation (WHO) performance status of 0 or 1 (Appendix 1)
7. Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week before the patient goes on study.

   Lab Test Value Required Haemoglobin (Hb) ≥9.0 g/dl Neutrophils ≥1.5 x 10^9/L Platelets (Plts) ≥100 x 10^9/L Serum bilirubin ≤1.5 x upper normal limit Alanine amino-transferase (ALT) and/or ≤ 2.5 x upper limit of normal (ULN) aspartate amino-transferase (AST) unless due to tumour in which case up to 5 x ULN is permissible Glomerular Filtration Rate (GFR) calculated either by the Wright formula ≥50 ml/min or Cockcroft-Gault formula or by isotope clearance measurement
8. 18 years or over
9. Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up

EXCLUSION CRITERIA

1. Radiotherapy (except for palliative reasons), endocrine therapy, immunotherapy, chemotherapy, biological agents or investigational agents during the previous 4 weeks (6 weeks for nitrosoureas and Mitomycin-C) before treatment.
2. Ongoing toxic manifestations of previous treatments. Exceptions to this are alopecia or certain Grade 1 toxicities, which in the opinion of the Investigator and the Drug Development Office (DDO) should not exclude the patient.
3. Known brain metastases.
4. Female patients able to become pregnant (or already pregnant or lactating). However, those female patients who have a negative serum or urine pregnancy test before enrolment and agree to use two highly effective forms of contraception (oral, injected or implanted hormonal contraception and condom, have an intrauterine device and condom, diaphragm with spermicidal gel and condom, or are surgically sterilised) 4 weeks before entering the trial, during the trial and for 6 months afterwards are considered eligible.
5. Male patients with partners of child-bearing potential (unless they agree to use one form of highly effective contraception such as a barrier method of condom plus spermicide during the trial and for 6 months afterwards).
6. Major thoracic and/or abdominal surgery in the preceding 4 weeks from which the patient has not recovered.
7. At high medical risk because of non-malignant systemic disease including active uncontrolled infection.
8. Concurrent malignancies at other sites, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin and concurrent breast and ovarian carcinoma. Cancer survivors, who have undergone potentially curative therapy for a prior malignancy, are eligible for the study.
9. Patients with active or unstable cardiac disease or history of myocardial infarction within 6 months. Patients with cardiovascular signs or symptoms should have a MUGA scan or echocardiogram, and those patients with left ventricular ejection fraction (LVEF) below the institutional limit of normal should be excluded.
10. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.
11. Patients who have already received a PARP inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2007-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Assessment of antitumor activity according to RECIST using tumor size measured clinically or radiologically with CT scan, MRI, plain x-ray, or other imaging techniques
Safety profile

SECONDARY OUTCOMES:
Time to progression and overall survival
Plasma levels measured by Liquid Chromatography/Mass Spectrometry/Mass Spectrometry
Poly(ADP-ribose) polymerase (PARP) activity measured ex vivo using validated assays
To determine the optimal oral dosing regimen, based on the assessment of antitumor activity and the safety profile

OTHER OUTCOMES:
TERTIARY OUTCOMES
  PARP expression using quantitative Western blotting immuno-assays
TERTIARY OUTCOMES
  Pharmacogenomics including CYP2D6 and CYP3A5 enzymes, drug transport proteins, as well as polymorphisms in the genes coding for the PARP enzymes themselves
TERTIARY OUTCOMES
  BRCA mutation status, PARP activity, and PARP expression in tumor biopsy samples (when possible)
TERTIARY OUTCOMES
  DNA repair enzyme status using immunohistochemical techniques in paraffin sections from original diagnostic biopsies/operative procedures (where available)
TERTIARY OUTCOMES
  DNA double strand break repair pathway function in cells obtained from ascitic or pleural fluid (where available) for primary cell culture and analysis for DNA repair

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Plummer, Principal Investigator — Northern Centre for Cancer Treatment at Newcastle General Hospital
Locations (7):
- United Kingdom (7):
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Cancer Research UK and University College London Cancer Trials Centre, London, England
  - Christie Hospital, Manchester, England
  - Sir Bobby Robson Cancer Trials Research Centre, Northern Centre for Cancer Care, Level 2, Freeman Hospital, Newcastle upon Tyne, England
  - Derriford Hospital, Plymouth, England
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland

REFERENCES:
- See also: Clinical Trial Results: A Cancer Research UK Phase II Proof of Principle Trial of the activity of the PARP-1 inhibitor, AG-014699 — https://www.clinicaltrialsregister.eu/ctr-search/trial/2006-002348-27/results